CLINICAL TRIAL: NCT01047137
Title: Effect of Psychological Stress Intervention on Chronic Urticaria Activity and Immune Dysregulation
Brief Title: Response of Urticaria to Stress Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled. A pilot study variation of this study was done instead.
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-0013
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2011-08

CONDITIONS: Chronic Urticaria
Keywords: Urticaria; Hives; Stress; Immune dysregulation
MeSH Terms: conditions — Chronic Urticaria; Urticaria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Participants will meet with a psychiatry resident once a week for six consecutive weeks for general supportive therapy, which will not provide psychological stress intervention.
  Interventions: Behavioral: General Supportive Therapy
- Intervention (Experimental): Participants will meet with a psychiatry resident once a week for six consecutive weeks to be educated on psychological stress intervention techniques.
  Interventions: Behavioral: Psychological Stress Intervention

INTERVENTIONS:
Behavioral: Psychological Stress Intervention — Intervention group participants will meet with a psychiatry resident once a week for six consecutive weeks to be educated on psychological stress intervention techniques focusing on relaxation, mindfulness, emotion regulation and acceptance and willingness.
  Arms: Intervention
Behavioral: General Supportive Therapy — There is no focus on stress intervention.
  Arms: Control

SUMMARY:
Several studies have shown a relationship between psychological stress and chronic urticaria (hives). The primary objective of this study is to evaluate the effect psychological stress intervention has on chronic urticaria.

DETAILED DESCRIPTION:
As many patients with chronic urticaria display heightened levels of stress before and/or after the onset of the urticaria, the purpose of this study is to evaluate the effect of psychological stress intervention on chronic urticaria. Intervention group participants will meet with a psychiatry resident once a week for six consecutive weeks to be educated on psychological stress intervention techniques. Control group participants will meet with a psychiatry resident once a week for six consecutive weeks for general supportive therapy, which will not provide psychological stress intervention. All participants will complete a packet of psychological and dermatological questionnaires before the first session with the psychiatry resident and one week after the final session. All participants will record daily 1) their urticaria symptoms and 2) the type and number of antihistamines taken. Blood and saliva samples will be collected before the first session and one week after completion of the final session to compare the levels of stress hormones and cytokines in order to evaluate an effect on immune dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-64 years who are inadequately controlled on H1 and/or H2-blocker therapy for chronic urticaria
* The Urticaria Activity Score must have a score of at least 2 (one point from each of the two categories: number of hives and severity of pruritus).

Exclusion Criteria:

* Urticaria secondary to vasculitis
* Use of prednisone, hydroxychloroquine, cyclosporine, or a tricyclic antidepressant (except Doxepin) within the 30 days prior to enrollment
* A history of anaphylaxis
* Non-controlled or debilitating chronic diseases (poorly controlled diabetes or congestive heart failure)
* An immune system disorder
* Deranged stress hormone level (for example, Cushing's disease)
* Ongoing omalizumab therapy
* Nocturnal employment (which would effect study measures, such as cortisol levels).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect psychological stress intervention has on chronic urticaria as measured by the Urticaria Activity Score | 6 weeks

SECONDARY OUTCOMES:
Comparison of the pre-intervention and post-intervention symptoms as determined by a packet of psychological and dermatological questionnaires. | 6 weeks
Evaluate pre- and post-intervention cytokine and stress hormone levels. | 6 weeks
The number of as-needed antihistamines used as the study progresses. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John W Tole, D.O., Principal Investigator — University of Mississippi Medical Center Div of Allergy and Immunology; Gailen D Marshall, M.D., Study Director — University of Mississippi Medical Center Div of Allergy and Immunology; Kim L Gratz, Ph.D., Study Director — University of Mississippi Medical Center Div of Psychiatry
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Mississippi, Jackson, Mississippi

REFERENCES:
- [Background] Powell RJ, Du Toit GL, Siddique N, Leech SC, Dixon TA, Clark AT, Mirakian R, Walker SM, Huber PA, Nasser SM; British Society for Allergy and Clinical Immunology (BSACI). BSACI guidelines for the management of chronic urticaria and angio-oedema. Clin Exp Allergy. 2007 May;37(5):631-50. doi: 10.1111/j.1365-2222.2007.02678.x. PMID 17456211
- [Background] Sperber J, Shaw J, Bruce S. Psychological components and the role of adjunct interventions in chronic idiopathic urticaria. Psychother Psychosom. 1989;51(3):135-41. doi: 10.1159/000288147. PMID 2636418
- [Background] Papadopoulou N, Kalogeromitros D, Staurianeas NG, Tiblalexi D, Theoharides TC. Corticotropin-releasing hormone receptor-1 and histidine decarboxylase expression in chronic urticaria. J Invest Dermatol. 2005 Nov;125(5):952-5. doi: 10.1111/j.0022-202X.2005.23913.x. PMID 16297195
- [Background] Yang HY, Sun CC, Wu YC, Wang JD. Stress, insomnia, and chronic idiopathic urticaria--a case-control study. J Formos Med Assoc. 2005 Apr;104(4):254-63. PMID 15909063
- [Background] Ozkan M, Oflaz SB, Kocaman N, Ozseker F, Gelincik A, Buyukozturk S, Ozkan S, Colakoglu B. Psychiatric morbidity and quality of life in patients with chronic idiopathic urticaria. Ann Allergy Asthma Immunol. 2007 Jul;99(1):29-33. doi: 10.1016/S1081-1206(10)60617-5. PMID 17650826
- [Background] Silvares MR, Coelho KI, Dalben I, Lastoria JC, Abbade LP. Sociodemographic and clinical characteristics, causal factors and evolution of a group of patients with chronic urticaria-angioedema. Sao Paulo Med J. 2007 Sep 6;125(5):281-5. doi: 10.1590/s1516-31802007000500006. PMID 18094895
- [Background] Berrino AM, Voltolini S, Fiaschi D, Pellegrini S, Bignardi D, Minale P, Troise C, Maura E. Chronic urticaria: importance of a medical-psychological approach. Eur Ann Allergy Clin Immunol. 2006 May;38(5):149-52. PMID 17058846
- [Background] Annesi-Maesano I, Beyer A, Marmouz F, Mathelier-Fusade P, Vervloet D, Bauchau V. Do patients with skin allergies have higher levels of anxiety than patients with allergic respiratory diseases? Results of a large-scale cross-sectional study in a French population. Br J Dermatol. 2006 Jun;154(6):1128-36. doi: 10.1111/j.1365-2133.2006.07186.x. PMID 16704645
- [Background] Marshall GD. Neuroendocrine mechanisms of immune dysregulation: applications to allergy and asthma. Ann Allergy Asthma Immunol. 2004 Aug;93(2 Suppl 1):S11-7. doi: 10.1016/s1081-1206(10)61482-2. PMID 15330008
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Zuberbier T, Bindslev-Jensen C, Canonica W, Grattan CE, Greaves MW, Henz BM, Kapp A, Kozel MM, Maurer M, Merk HF, Schafer T, Simon D, Vena GA, Wedi B; EAACI/GA2LEN/EDF. EAACI/GA2LEN/EDF guideline: definition, classification and diagnosis of urticaria. Allergy. 2006 Mar;61(3):316-20. doi: 10.1111/j.1398-9995.2005.00964.x. PMID 16436140